CLINICAL TRIAL: NCT00947180
Title: Randomized Controlled Trial Comparing Biofeedback, Electrogalvanic Stimulation, and Massage for the Treatment of Chronic Proctalgia
Brief Title: Gastrointestinal Biopsychosocial Research Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R24 DK67674 (completed); R24DK067674 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-07-27 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2010-03

CONDITIONS: Chronic Proctalgia (Also Called Levator Ani Syndrome)
Keywords: Biofeedback; Pelvic floor; Levator ani syndrome; Chronic proctalgia; Electrogalvanic stimulation; Massage
MeSH Terms: conditions — Levator syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrogalvanic stimulation (Active Comparator): High voltage electrical stimulation was delivered through an anal plug to induce relaxation of pelvic floor muscles.
  Interventions: Other: Electrogalvanic stimulation
- Digital massage (Active Comparator): The therapist massaged the levator ani muscles by applying firm pressure with a gloved finger and rotating from left to right.
  Interventions: Behavioral: Digital massage
- Biofeedback (Experimental): Electromyographic (EMG) activity was recorded from a probe in the anal canal, averaged and displayed to patients to help them learn to relax pelvic floor muscles during straining.
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback — Electromyographic (EMG) activity was recorded from sensors placed in the anal canal, averaged, and displayed to patients to help them learn to relax the pelvic floor muscles during straining.
  Arms: Biofeedback
Other: Electrogalvanic stimulation — Electrical stimulation was applied to pelvic floor muscles through an anal plug. Frequency was 80 pulses per sec, and voltage was slowly increased from 0 to 150-350 volts as tolerated.
  Arms: Electrogalvanic stimulation
Behavioral: Digital massage — Using a gloved finger, the therapist pressed on the levator ani as firmly as tolerated and moved the finger from side to side 3-4 times.
  Arms: Digital massage

SUMMARY:
This study has been completed. The following is a brief description of the aims, methods, and results of the study:

Previous small studies suggest that chronic proctalgia (chronic recurring pain in the anal canal or rectum), which is also called levator ani syndrome, can be treated with biofeedback to teach relaxation of pelvic floor muscles, or electrogalvanic stimulation (electrical stimulation to relax muscles), or massage of pelvic floor muscles. The aim of this study was to compare the effectiveness of these three treatments, to determine how they work physiologically, and to identify which patients are most likely to benefit.

Methods: Subjects had to meet the diagnostic criteria for chronic proctalgia and to report pain at least once a week. They had to also be free of medical or psychiatric disorders that could explain their chronic proctalgia. Patients qualified to enter the study were separated into two groups based on whether they reported tenderness when the examining physician pressed on the levator ani muscles of the pelvic floor. All 157 patients who were enrolled received 9 sessions of psychological counseling plus biofeedback or electrogalvanic stimulation or massage. The results of treatment were assessed at 1, 3, 6, and 12 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria: Recurring episodes of pain or aching in the anal canal or rectum for at least 12 weeks in the previous year. Episodes last at least 20 minutes. Pain must occur at least weekly during a 4-week run-in.

Exclusion Criteria: Other medical or psychiatric diagnoses that could explain recurring rectal pain. Daily use of psychotropic medications. Meets diagnostic criteria for irritable bowel syndrome or functional constipation. Screening studies included physical examination by a gastroenterologist, colonoscopy, pelvic ultrasound, and surgical consult in all patients and referral to a gynecologist or urologist if indicated by history.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2000-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adequate relief of pain (proctalgia) | 1, 3, 6, and 12 months following treatment

SECONDARY OUTCOMES:
Subjective pain improvement (ordinal scale) | 1, 3, and 6 months follow-up
Number of days per month with rectal pain (inferred from 30 day symptom diary) | Baseline, then 1, 3, and 6 months follow-up
Visual analog scale rating of pain averaged across weeks for 30 day diary period | Baseline, then 1, 3, and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Division of Gastroenterology at the University of Verona, Verona, Italy

REFERENCES:
- [Result] Chiarioni G, Nardo A, Vantini I, Romito A, Whitehead WE. Biofeedback is superior to electrogalvanic stimulation and massage for treatment of levator ani syndrome. Gastroenterology. 2010 Apr;138(4):1321-9. doi: 10.1053/j.gastro.2009.12.040. Epub 2010 Jan 4. PMID 20044997